CLINICAL TRIAL: NCT05415527
Title: Evaluation of Pretreatment Sarcopenia in Patients With Inoperable High-grade Ovarian Carcinoma as Part of Optimised Management
Acronym: OPTIMOVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IB2021-05
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Carcinoma
Keywords: Inoperable high-grade ovarian carcinoma; Sarcopenia evaluation; nutritional monitoring; adapted physical activity
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Glutamyl Aminopeptidase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with inoperable high-grade ovarian carcinoma (Other): Evaluation of sarcopenia in patients with inoperable high-grade ovarian carcinoma as part of optimised management
  Interventions: Other: Presence of sarcopenia evaluated prior to neoadjuvant chemotherapy and during chemotherapy as part of optimised management(dietician and APA).

INTERVENTIONS:
Other: Presence of sarcopenia evaluated prior to neoadjuvant chemotherapy and during chemotherapy as part of optimised management(dietician and APA). — Sarcopenia will be evaluated by CT-scan. This method will be combined with a bone mineral density test which is also a way of entering into a more specific approach to sarcopenia screening.
  The patients will receive optimised treatment by nutritional monitoring and adapted physical activity (APA) in addition to follow-up for sarcopenia.

SUMMARY:
Prospective, monocentric study evaluating the presence of sarcopenia prior to neoadjuvant chemotherapy and during chemotherapy as part of optimised management.

DETAILED DESCRIPTION:
Prior to carrying out the research, the informed consent of the person must be obtained after being informed of the purpose of the research, its conduct and duration, benefits, potential risks and constraints of the study.

Before inclusion,all eligibility criteria will be verified.

Sarcopenia in patients with inoperable, high-grade epithelial ovarian carcinoma will be evaluated at different times:

* before treatment, in the 30 days prior to their inclusion in the study,
* after 3 neoadjuvant chemotherapy cycles,
* after 3 adjuvant chemotherapy cycles,
* 9 months after surgery. The reference detection method is by CT-scan. This will be combined with a bone mineral density test which is also a way of entering into a more specific approach to sarcopenia screening.

On inclusion, the patients will receive optimised treatment by nutritional monitoring and adapted physical activity (APA) in addition to follow-up for sarcopenia.

This follow-up by a dietician and a physical fitness trainer will be recorded at each neoadjuvant chemotherapy session.

Dietary advice will be given each time along with personalised advice if weight loss were to be observed.

If undernutrition or a foreseeable risk of undernutrition are diagnosed, parenteral nutrition will be prescribed by the oncologist, the anaesthetist or the surgeon.

The objective of APA is to prevent the onset or aggravation of disease, to increase patient autonomy and quality-of-life, or even to help them return to social activities.

Respiratory preparation will also be offered to increase the patient's respiratory capacity in view of surgery, with exercises to be done using a respiratory training device.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Inoperable, high-grade, epithelial ovarian carcinoma requiring perioperative chemotherapy (neoadjuvant and adjuvant).
3. Optical medical treatment (carboplatin-taxol chemotherapy every 3 weeks) and surgery at Institut Bergonié.
4. Non-clinically undernourished patient, i.e. without loss of more than 10% bodyweight in 6 months
5. Free, informed and written consent signed by the participant and the investigator (on the day of inclusion at the latest and before any tests required for the research).
6. Patient with social security cover in accordance with Article 1121-11 of the French code of public health.

Exclusion Criteria:

1. Contraindication to CT-scans.
2. Contraindication to bone mineral densitometry.
3. Patients over the age of 70 the G8 of whom requires oncogeriatric surgery.
4. Patients under guardianship, vulnerable patients or patients under any other legal protection measures.
5. Geographic, social or psychological factors meaning the patient is unable to commit to study follow-up and procedures.
6. Patient already included in this study or in another study evaluating the impact of sarcopenia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2027-06-10 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with pretreatment sarcopenia identified by analysis of the baseline CT-scan (CT0). | Baseline
  Proportion of patients with pretreatment sarcopenia identified by analysis of the baseline CT-scan (CT0). According to the 2019 HAS guidelines [Diagnosis of undernutrition in children and adults, November 2019], we consider the patient to have sarcopenia if her MSI is strictly below 38.5 cm2/m2.

SECONDARY OUTCOMES:
The time of access to chemotherapy | From the date of surgery to the start date of adjuvant chemotherapy, assessed up to 2 months from surgery
  The time of access to chemotherapy is the time between the date of surgery and the adjuvant chemotherapy start date. Pretreatment sarcopenia is defined as for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre GEKIERE, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, France